CLINICAL TRIAL: NCT05698381
Title: Effect of Daily Vinegar Ingestion for Four Weeks on Mood State, Inflammatory State, and Risk for Metabolic Syndrome in Healthy Adults
Brief Title: Daily Vinegar Ingestion and Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Associate Dean, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00017204
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Inflammation; Metabolic Syndrome; Depression
Keywords: vinegar; acetic acid; LPS
MeSH Terms: conditions — Inflammation; Metabolic Syndrome; Depression | interventions — Acetic Acid

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: liquid vinegar (contains active dose of acetic acid) vinegar pill (contains only a trace of acetic acid)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid vinegar (Experimental): 4 tablespoons BID per day (3000 mg acetic acid)
  Interventions: Dietary Supplement: Liquid vinegar
- Vinegar pill (Placebo Comparator): 2 vinegar pills per day (30 mg acetic acid)
  Interventions: Dietary Supplement: Vinegar pill

INTERVENTIONS:
Dietary Supplement: Liquid vinegar — 2 tablespoons consumed twice daily with meals
  Arms: Liquid vinegar
Dietary Supplement: Vinegar pill — 2 pills consumed upon waking
  Arms: Vinegar pill

SUMMARY:
The purpose of this study is to determine if vinegar ingestion promotes beneficial changes to metabolic health parameters in healthy, overweight adults.

DETAILED DESCRIPTION:
Recent research, in animal and human subjects, suggests that vinegar intake is inversely associated with insulin resistance, mood states and depression, inflammation, and other disease parameters. The study will be conducted as a randomized controlled trial in overweight adults to further examine these relationships and possible mechanisms. Although the mechanisms are not known, research suggests that changes in the gut microbiome, a response to the ingestion of the postbiotic acetic acid, may factor into the beneficial effects of vinegar ingestion. Through analyses of blood, changes in key blood metabolites associated with mood states (e.g., gamma-aminobutyric acid) as well as markers of gut health (e.g., LPS binding protein) and inflammation (e.g., CRP) will be assessed. Additionally mood state will be assessed using validated measures and determine risk for metabolic syndrome, a cluster of risk factors associated with many chronic conditions. It is hypothesized that vinegar ingestion will promote beneficial changes to these health parameters.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoker
* free of chronic disease by self-report
* able to speak, read, and understand English
* able to consent.
* BMI ≥ 25 and ≤ 35

Exclusion Criteria:

* adherence to specific diets for weight loss
* vegetarian
* report GERD or regular heartburn
* unwilling to consume vinegar daily for 4 weeks
* pregnant or lactating women
* recreational drug use, alcohol intake above recommendations (1 drink/day for women, 2 drinks/day for men - or none)
* competitive level physical training (e.g., physical activity above recommendations as set by the Physical Activity Guidelines for Americans)
* scoring 1 or higher on question 9 of the PHQ-9 questionnaire.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Depression score | change from baseline at week 4
  Patient Health Questionnaire (PHQ-9); scores range from 0 (none-minimal) to 27 (severe)
Depression score | change from baseline at week 4
  Center for Epidemiologic Studies Depression Scale (CES-D); scores range from 0 to 60 (higher scores suggest a greater presence of depressive symptoms. A score of 15 or higher is interpreted to indicate a risk for depression).
gamma-aminobutyric acid (GABA) | change from baseline at week 4
  Blood levels of the neurotransmitter GABA

SECONDARY OUTCOMES:
metabolic syndrome | change from baseline at week 4
  A cluster of conditions that increase risk of heart disease, stroke and type 2 diabetes: increased blood pressure, high blood sugar, waist circumference, and abnormal cholesterol or triglyceride levels. siMS score = 2*Waist/Height + Gly/5.6 + Tg/1.7 + TAsystolic/130-HDL/1.02 or 1.28 (for male or female subjects, respectively) (adapted from Soldatovic et al. (2016) siMS Score: Simple Method for Quantifying Metabolic Syndrome. PLoS ONE 11(1): e014614)
Inflammation | change from baseline at week 4
  Blood C-reactive protein
LPS | change from baseline at week 4
  Blood Lipopolysaccharide binding protein

CONTACTS AND LOCATIONS:
Overall Officials: Carol S Johnston, PhD, Principal Investigator — Arizona State University
Locations (1):
- 850 PBC, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No